CLINICAL TRIAL: NCT05591534
Title: Endorectal Brachytherapy for Dose Escalation in Rectal Preservation Treatment of Rectal Cancer (ICUREC)
Brief Title: Endorectal Brachytherapy for Rectal Cancer
Acronym: ICUREC
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Unknown time frame for availability of new endorectal probes
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2021/38
Record Dates: First submitted 2022-10-11; First posted 2022-10-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Rectal Carcinoma
Keywords: Endorectal brachytherapy; Rectal cancer; Radiotherapy; Non-operative management
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endorectal brachytherapy (Experimental): Endorectal brachytherapy
  Interventions: Radiation: Endorectal brachytherapy

INTERVENTIONS:
Radiation: Endorectal brachytherapy — Endorectal brachytherapy : 30 Gy in 3 sessions of 10 Gy delivered weekly

SUMMARY:
The management of rectal cancers has changed over the past decades towards a multidisciplinary strategy, combining radiotherapy, chemotherapy, and surgery. Local recurrence rates, dropped to less than 6 % with pre-operative radiotherapy and the standardization of total mesorectal excision (TME), at the price of increased peri-operative morbidity and functional sequelae. Since neoadjuvant treatment achieves up to 30 % complete response, organ preservation has been increasingly debated for good responders. With the introduction of better-quality imaging for tumour visualization and treatment planning, a new targeted radiation treatment was introduced with high dose rate endorectal brachytherapy (HDRBT), developped by Dr Te Vuong's team in Montreal. This treatment allows for radiotherapy dose escalation to increase the complete response rate, and subsequently the rate of patients amenable to rectal preservation. This phase 2 trial study is proposed to assess the feasibility of HDR brachytherapy after standard chemoradiotherapy among patients selected for rectal preservation.

DETAILED DESCRIPTION:
The standard treatment for locally advanced rectal cancer consists in chemoradiotherapy followed by radical surgery with total mesorectal excision (TME) and adjuvant chemotherapy depending on lymph node status. This radiosurgical strategy has reduced local recurrence rates to less than 5% in expert centers, but at the cost of 20-30% morbidity and functional sequelae. Chemoradiotherapy can sterilize 15% of tumors, and up to 30% when neoadjuvant chemotherapy is given, calling into question the usefulness of systematic radical surgery in good responders. Ongoing trials are looking at treatment intensification either by chemotherapy intensification or by dose escalation in radiotherapy, with the aim of increasing the rectal preservation rate. Endorectal brachytherapy, developed by Prof. Té Vuong in Montreal, makes it possible to deliver a complementary dose directly to the tumor using a high-activity Iridium-192 radioactive source. It is an ambulatory treatment, which allows to deliver a complementary dose of 30 Gy in 3 sessions of 10 Gy at one week interval after external radiotherapy.

The objective of our trial is to demonstrate the feasibility of rectal brachytherapy for our patients in France with an acceptable toxicity rate similar to that described by the Canadian teams. In addition, this bicentric trial will allow to prove capacity to train radiotherapist colleagues in the technique of endorectal brachytherapy, which is an essential prerequisite for the development of the technique throughout France.

Main objective : To assess the feasibility of endorectal brachytherapy in patients showing partial response after standard neoadjuvant therapy with a goal of rectal preservation.

Secondary objectives: To describe the potential efficacy of endorectal brachytherapy in patients with partial response after standard neoadjuvant therapy by the complete clinical response rate and complete radiological response rate on MRI at 8 weeks, 4 months, 8 months, and 1 year, local recurrence rate, recurrence-free survival, and overall survival at 1 year Describe the rate of curative surgery (R0) in case of recurrence as well as the surgical morbidity according to the Dindo-Clavien score at 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven rectal adenocarcinoma
* Tumor cT2T3Tumor N0 or N1, M0
* Size < 6cm and < 50% of circumference at initial workup, location ≤ 10 cm from anal margin
* Partial response assessed on MRI 3-8 weeks after completion of external beam radiation therapy
* Resolved rectal toxicity from external radiotherapy (grade ≤ 1) at the time of inclusion
* ECOG performance index ≤ 2
* Patient ≥ 18 years of age
* Patient likely to receive radiation therapy
* Effective contraception for patients of childbearing potential: male patients and women of childbearing potential must agree to use two medically validated methods of contraception (one for the patient and one for the partner) during treatment and at least until 6 months after the last treatment
* Informing the patient and obtaining free, informed and written consent, signed by the patient and the investigator
* Subject affiliated or beneficiary of a social security system of a member state of the European Community (article L1121-11 of the Public Health Code)

Exclusion Criteria:

* T1 or T4 tumor
* Tumor size > 6 cm or > 50% of circumference at initial workup
* Invaded external sphincter or levator ani
* N2 tumor (> 3 positive nodes)
* Upper rectal tumor (> 10 cm from anal margin)
* Metastatic disease
* Contraindication to radiotherapy
* Unusual and unresolved rectal toxicity from external radiation therapy (> grade 1) at the time of inclusion
* Pregnant, potentially pregnant, or breastfeeding women
* Persons deprived of liberty or under guardianship or unable to give consent
* Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Tolerance | 8 weeks after the end of treatment
  Proportion of patients receiving the 3 brachytherapy sessions without acute grade 3 proctitis (requiring hospitalization or transfusion) within 8 weeks after the end of treatment

SECONDARY OUTCOMES:
Complete clinical response | At 8 weeks, 4 months, 8 months and 1 year
  Proportion of patients with a complete clinical response
Complete radiological response | At 8 weeks, 4 months, 8 months and 1 year
  Proportion of patients with a complete radiological response on MRI
Local recurrence | At 1 year
  Proportion of patients with a local recurrence up to 1 year
Recurrence-free survival | At 1 year
Overall survival | At 1 year
Quality of life (EORTC QLQ C30) | At 8 weeks, 4 months, 8 months and 1 year
  The scores of questionnaire QLQ C-30 will be examined. The EORTC QLQ-C30 is a patients self-rating questionnaire that measures physical, role, social, emotional, and cognitive functions as well as overall QoL. Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales
Quality of life (EORTC QLQ CR29) | At 8 weeks, 4 months, 8 months and 1 year
  The scores of questionnaire QLQ CR-29 will be examined. The EORTC QLQ-CR29 has five functional and 18 symptom scales. Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales
Low Anterior Resection Syndrome score (LARS score) | At 8 weeks, 4 months, 8 months and 1 year
  The LARS questionnaire (low anterior resection score) evaluates bowel function. Five questions regarding incontinence for flatus and liquid stools, frequency, clustering and urgency for defecation are taken into account. The score ranges from 0 to 42 is divides into no LARS (0 to 20 points), minor LARS (21 to 29 points), and major LARS (30 to 42 points)
Curative surgery for recurrence | Up to 1 year
  Proportion of curative surgery in case of recurrence (R0)
Surgical morbidity for recurrence | 3 months after surgery
  Proportion of patients with and description of surgical morbidity (Dindo) at 3 months in case of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Véronique VENDRELY, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux, Service de Radiothérapie, Bordeaux
  - APHP - Hôpital Tenon, Service Oncologie-Radiothérapie, Paris

IPD SHARING:
Plan to Share IPD: No